CLINICAL TRIAL: NCT04247919
Title: Investigation of Genetic Variations on Patients With Adverse Drug Events While on Direct Oral Anticoagulants (DOACs)
Brief Title: DOAC ADRs Retrospective Study
Status: Terminated | Type: Observational
Why Stopped: Limitations to recruitment due to COVID-19
Sponsor: Cipherome, Inc. (Industry)
Collaborators: Santa Clara Valley Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: C02-001 SC002
Record Dates: First submitted 2020-01-22; First posted 2020-01-30 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Drug-Related Side Effects and Adverse Reactions
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Study participants will either submit saliva samples or have a laboratory drawn blood sample.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study's objective is to evaluate if Cipherome's algorithm could have predicted the serious adverse drug reactions (ADRs) experienced by patients while on direct oral anti-coagulants (DOACs).

DETAILED DESCRIPTION:
Using the latest next generation sequencing tools, this study will evaluate adverse drug reactions (ADRs) (e.g., major bleeding or treatment failure) in study participants while on direct oral anticoagulants (DOACs). A web-based program will analyze the data obtain from sequencing, and generate a drug safety score (DSS). The DSS risk score will be compared with pre-specified serious ADRs associated with DOAC therapy. A secondary analysis will involve discovery of novel variants that arise from our analysis and may potentially affect the outcome of DOAC treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient 18 years and older, who experienced a serious adverse drug reaction while taking a DOAC and is able to provide informed consent.

Exclusion Criteria:

* Failure to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients on rivaroxaban, apixaban, and dabigatran who experienced a serious adverse drug reaction and/or treatment failure.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants with a Major Bleeding Event | Within 90 days of DOAC therapy initiation
  Reduction in hemoglobin of at least 2 g/dL Blood loss requiring transfusion of at least 2 units of whole blood or erythrocytes Critical anatomical sites of bleeding: intramuscular with compartment syndrome, intracranial, intraspinal, retroperitoneal, intraocular, pericardial, and atraumatic intra-articular bleeding.
  Bleeding led to death
Number of Participants with a Clinically Relevant Non-major Bleeding Event | Within 90 days of DOAC therapy initiation
  Acute or subacute clinically overt bleed that does not meet the criteria for a major bleed but prompts a clinical response, in that it leads to at least one of the following:
  A hospital admission for bleeding, or A physician guided medical or surgical treatment for bleeding, or A change in antithrombotic therapy (including interruption or discontinuation of study drug).
Number of Deaths Reported | Through study completion, an average of 1 year
  Death at any time

SECONDARY OUTCOMES:
Number of Participants with a Thromboembolic Event | Within 90 days of DOAC therapy initiation
  Deep vein thrombosis, pulmonary embolism, ischemic stroke, transient ischemic attack, arterial thrombosis, or other thromboembolic event.

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Wang, MD, Principal Investigator — Santa Clara Valley Medical Center; Michelle Wilson, MD, Study Director — Santa Clara Valley Medical Center; Jessica Song, PharmD, Study Director — Santa Clara Valley Medical Center
Locations (1):
- Santa Clara Valley Medical Center, San Jose, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colilla S, Crow A, Petkun W, Singer DE, Simon T, Liu X. Estimates of current and future incidence and prevalence of atrial fibrillation in the U.S. adult population. Am J Cardiol. 2013 Oct 15;112(8):1142-7. doi: 10.1016/j.amjcard.2013.05.063. Epub 2013 Jul 4. PMID 23831166
- [Background] Wysowski DK, Nourjah P, Swartz L. Bleeding complications with warfarin use: a prevalent adverse effect resulting in regulatory action. Arch Intern Med. 2007 Jul 9;167(13):1414-9. doi: 10.1001/archinte.167.13.1414. PMID 17620536
- [Background] Zareh M, Davis A, Henderson S. Reversal of warfarin-induced hemorrhage in the emergency department. West J Emerg Med. 2011 Nov;12(4):386-92. doi: 10.5811/westjem.2011.3.2051. PMID 22224125
- [Background] Kirley K, Qato DM, Kornfield R, Stafford RS, Alexander GC. National trends in oral anticoagulant use in the United States, 2007 to 2011. Circ Cardiovasc Qual Outcomes. 2012 Sep 1;5(5):615-21. doi: 10.1161/CIRCOUTCOMES.112.967299. Epub 2012 Sep 4. PMID 22949490
- [Background] Bauer KA. Pros and cons of new oral anticoagulants. Hematology Am Soc Hematol Educ Program. 2013;2013:464-70. doi: 10.1182/asheducation-2013.1.464. PMID 24319220
- [Background] Kanuri SH, Kreutz RP. Pharmacogenomics of Novel Direct Oral Anticoagulants: Newly Identified Genes and Genetic Variants. J Pers Med. 2019 Jan 17;9(1):7. doi: 10.3390/jpm9010007. PMID 30658513
- [Background] Sennesael AL, Larock AS, Douxfils J, Elens L, Stillemans G, Wiesen M, Taubert M, Dogne JM, Spinewine A, Mullier F. Rivaroxaban plasma levels in patients admitted for bleeding events: insights from a prospective study. Thromb J. 2018 Nov 12;16:28. doi: 10.1186/s12959-018-0183-3. eCollection 2018. PMID 30455596
- [Background] Ing Lorenzini K, Daali Y, Fontana P, Desmeules J, Samer C. Rivaroxaban-Induced Hemorrhage Associated with ABCB1 Genetic Defect. Front Pharmacol. 2016 Dec 19;7:494. doi: 10.3389/fphar.2016.00494. eCollection 2016. PMID 28066243
- [Background] Ueshima S, Hira D, Kimura Y, Fujii R, Tomitsuka C, Yamane T, Tabuchi Y, Ozawa T, Itoh H, Ohno S, Horie M, Terada T, Katsura T. Population pharmacokinetics and pharmacogenomics of apixaban in Japanese adult patients with atrial fibrillation. Br J Clin Pharmacol. 2018 Jun;84(6):1301-1312. doi: 10.1111/bcp.13561. Epub 2018 Apr 16. PMID 29457840
- [Background] Shi J, Wang X, Nguyen JH, Bleske BE, Liang Y, Liu L, Zhu HJ. Dabigatran etexilate activation is affected by the CES1 genetic polymorphism G143E (rs71647871) and gender. Biochem Pharmacol. 2016 Nov 1;119:76-84. doi: 10.1016/j.bcp.2016.09.003. Epub 2016 Sep 8. PMID 27614009
- [Background] Dimatteo C, D'Andrea G, Vecchione G, Paoletti O, Cappucci F, Tiscia GL, Buono M, Grandone E, Testa S, Margaglione M. Pharmacogenetics of dabigatran etexilate interindividual variability. Thromb Res. 2016 Aug;144:1-5. doi: 10.1016/j.thromres.2016.05.025. Epub 2016 May 26. PMID 27261537
- [Background] Sychev DA, Levanov AN, Shelekhova TV, Bochkov PO, Denisenko NP, Ryzhikova KA, Mirzaev KB, Grishina EA, Gavrilov MA, Ramenskaya GV, Kozlov AV, Bogoslovsky T. The impact of ABCB1 (rs1045642 and rs4148738) and CES1 (rs2244613) gene polymorphisms on dabigatran equilibrium peak concentration in patients after total knee arthroplasty. Pharmgenomics Pers Med. 2018 Jul 25;11:127-137. doi: 10.2147/PGPM.S169277. eCollection 2018. PMID 30100750
- [Background] 1000 Genomes Project Consortium; Auton A, Brooks LD, Durbin RM, Garrison EP, Kang HM, Korbel JO, Marchini JL, McCarthy S, McVean GA, Abecasis GR. A global reference for human genetic variation. Nature. 2015 Oct 1;526(7571):68-74. doi: 10.1038/nature15393. PMID 26432245